CLINICAL TRIAL: NCT03603821
Title: Quantitative Comparison of Results Obtained by Self-administered IPSS, Sanitary Staff-supervised IPSS and Directed Medical History and Its Correlation With Clinical Parameters in the Assessment of Lower Urinary Tract Symptoms in Males
Brief Title: Comparison of Self-administered IPSS, Sanitary Staff-supervised IPSS, Medical History and Clinical Parameters
Acronym: KILL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, EDUARDO VICENTE PALACIO, Senior and Consultor Staff in the Department of Urology, Corporacion Parc Tauli
Other Study IDs: Kill IPSS
Record Dates: First submitted 2018-07-16; First posted 2018-07-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: LUTS; QUESTIONNAIRE; IPSS
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUTS male: Clinical assesment of males older than 50 years with lower urinary tract symptoms presumably related to benign prostate enlargement
  Interventions: Diagnostic Test: CLINICAL ASSESMENT

INTERVENTIONS:
Diagnostic Test: CLINICAL ASSESMENT — IPSS questionnaire, uroflowmetry, prostate and bladder ultrasonography, voiding diary, medical interview
  Other Names: Ultrasonography; IPSS questionnaire; Voiding diary; Uroflowmetry

SUMMARY:
Descriptive prospective study carried out to compare the results obtained by self-administered IPSS (International Prostate Symptom Score), Sanitary staff-supervised IPSS and directed medical interview and its correlation with clinical parameters in the assessment of lower urinary tract symptoms in males.

DETAILED DESCRIPTION:
The IPSS is a validated questionnaire (also in spanish language) widely used to evaluate lower urinary tract symptoms (LUTS) in males. It contains 7 multiple-choice questions related to urinary symptoms with a Likert response scale and 1 question assessing quality of life. This test has been approved for self-administration and its purpose is quantifying and monitoring symptoms severity.

The aim of this study is to compare the scores achieved in a self-administered IPSS questionnaire with those obtained when the questionnaire is answered with the help and supervision of a sanitary staff. These results will also be contrasted with the scores retrieved in a standard directed medical interview and correlated with objective functional parameters of lower urinary tract symptoms.

A descriptive prospective study will be carried out analysing lower urinary tract symptoms from patients over 50 years old.

All patients will be provided with a IPSS to be fulfilled at home and after a short period of time without any change in his LUTS treatment, the patient will repeat the questionnaire in the hospital under the supervision of a sanitary staff.

A standard structured medical interview focusing in LUTS will be performed to every patient. In order to compare the results achieved with both IPSS with those obtained during the interview a Likert score was assigned to each question.

At the same time, objective lower urinary tract symptoms data will be collected and compared to the results obtained previously with both the questionnaires and the medical interview. Uroflowmetry and post physiological void residual volume measurement with ultrasonography will be performed as evaluation of voiding symptoms. On the other hand, filling symptoms will be evaluated with a validated 3-day voiding diary to be accomplished previously to the medical visit.

Data to be collected includes Uroflowmetry parameters Qmax, Qm, curve shape type and time to Qmax, ultrasonographic PVR (post-void residual) measurement and daytime and nightime number of voids, medium volume of void, number of urgency and urge incontinence episodes and maximal vesical functional volume wich will be extracted from the 3-day voiding diary.

A statistical analysis will be performed to compare the scores obtained through the questionnaires and the medical interview and the correlation of each of them with the objective clinical parameters obtained.

ELIGIBILITY:
Inclusion Criteria:

* males older than 50 years, with LUTS

Exclusion Criteria:

* Urinary tract infection
* Bladder tumor o lithiasis
* changes in LUTS treatment during the analysis period (pharmacological or surgical)
* urethral manipulation during the analysis period (catheterization or cystoscopy)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males older than 50 years with low urinary symptoms followed in the investigator's Urology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
correlation between different clinical severity scores in LUTS | data will be measured once all questionnaires are provided and objective explorations performed. All data will be obtained in a maximum of 30 days period for each patient. During this period of time the patient will not change any of his treatments.
  correlation between the scores obtained with an self-administered IPSS, a sanitary staff-supervised IPSS and a standard medical interview focused on LUTS based on a Likert severity scale 0-4 (5 levels of severity)

SECONDARY OUTCOMES:
correlation between clinical severity scores and objective severity symptoms | data will be measured once all questionnaires are provided and objective explorations performed. All data will be obtained in a maximum of 30 days period for each patient. During this period of time the patient will not change any of his treatments.
  correlation between the scores obtained with IPSS (self-administered and nurse-supervised and a standard medical interview with different objective clinical parameters of storage and voiding symptoms

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO VICENTE PALACIO, UROLOGIST, Study Director — CORPORATION PARC TAULI
Locations (1):
- Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes